CLINICAL TRIAL: NCT00876057
Title: Subtotal Versus Total Abdominal Hysterectomy- a Prospective Randomised Comparison of Medical , Psychological and Sexual Effects.
Brief Title: Psychological Well-being, Recovery and Sexuality After Total and Subtotal Hysterectomy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Linkoeping (Other)
Responsible Party: Principal Investigator, Preben Kjolhede, Professor, University Hospital, Linkoeping
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2009-0102
Record Dates: First submitted 2009-04-03; First posted 2009-04-06 (Estimated); Last update posted 2012-06-11 (Estimated); Status verified 2012-06

CONDITIONS: Hysterectomy
Keywords: psychological well-being; recovery; time in hospital; sick-leave; complications; Sexual well-being
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- TH (Active Comparator): Total hysterectomy
  Interventions: Procedure: Total abdominal hysterectomy
- SH (Active Comparator): Subtotal hysterectomy
  Interventions: Procedure: Subtotal abdominal hysterectomy

INTERVENTIONS:
Procedure: Total abdominal hysterectomy — Total abdominal hysterectomy
  Arms: TH
Procedure: Subtotal abdominal hysterectomy — Subtotal abdominal hysterectomy
  Arms: SH

SUMMARY:
The purpose of this study is to determine whether psychological well-being, recovery and sexuality differs in women undergoing subtotal and total abdominal hysterectomy.

Se also Detailed Description for additional study.

DETAILED DESCRIPTION:
An additional study study based on the material in original study started in april 2011. The purpose of this study is to investigate the development of pelvis organ prolapse in the long term (median eleven years after hysterectomy and by questionnaires, Pelvic-floor Distress Inventory SF-20 analyze if patient reported symptoms regarding urinary-and bowels functions differs regarding the method of hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

* Primarily uterine fibroids with bleeding disturbance or mechanical symptoms but other benign disorders were hysterectomy was recommended were also eligible
* After surgery at least one ovary preserved.
* Informed verbal and written consent
* Proficiency in Swedish

Exclusion Criteria:

* Malignancy in the genital organs.
* Previous or present cervical dysplasia.
* Rapidly growing fibroids where malignancy could not be ruled out
* Preoperative treatment with GnRH analogues.
* Postmenopausal women without hormone therapy
* Severe psychiatric disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 1998-03; Primary Completion 2004-04 (Actual); Study Completion 2005-04 (Actual)

PRIMARY OUTCOMES:
Psychological well-being | One year after surgery

SECONDARY OUTCOMES:
Recovery of general well-being | Five weeks after surgery
Sexuality | One year
Pelvic organ prolapse (anatomical) | 7-14 years
  Follow-up median eleven years after the initial hysterectomy. Clinical investigation including POP-Q.
Patient reported symptoms of pelvic organ dysfunction | 7-14 years
  Follow-up median eleven years after the initial hysterectomy. Questionnaire (Pelvic Floor Dysfuntion Inventoy).

CONTACTS AND LOCATIONS:
Overall Officials: Preben Kjölhede, MD, PhD, Study Chair — University Hospital, Linköping; Pär Persson, MD, Study Director — University Hospital, Linköping
Locations (7):
- Sweden (7):
  - Höglandssjukhuset i Eksjö, Eksjö
  - Ryhov Central Hospital, Jönköping
  - County Hospital in Kalmar, Kalmar
  - Motala Counbty Hospital, Motala
  - Vrinnevi Hospital, Norrköping
  - Capio Läkargruppen, Örebro
  - Värnamo County Hospital, Värnamo